CLINICAL TRIAL: NCT03616379
Title: Behavioral Strategies to Reduce Stress Reactivity in Opioid Use Disorder
Brief Title: Stress Response in Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, McHugh, R. Kathryn, Assistant Professor, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018P001419
Record Dates: First submitted 2018-07-05; First posted 2018-08-06 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The study PI and data analyst will be blind to study condition. The experimenter will and participant will be aware of the study condition because this is a behavioral intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psychoeducational Control (Placebo Comparator)
  Interventions: Behavioral: Psychoeducational Control
- Affect Regulation Condition (Experimental)
  Interventions: Behavioral: Affect Regulation
- Affect Labelling Condition (Experimental)
  Interventions: Behavioral: Affect Labelling

INTERVENTIONS:
Behavioral: Psychoeducational Control — The Psychoeducational Control condition will consist of a brief script describing the body's response to stress and will not discuss cognition or the role of interpretation or affect labeling during stress.
  Arms: Psychoeducational Control
Behavioral: Affect Regulation — In the Affect Regulation Condition, participants will be provided instructions for how to reappraise negative thoughts in the context of stress by developing statements consistent with more benign interpretations of stress (e.g., This won't last forever.).
  Arms: Affect Regulation Condition
Behavioral: Affect Labelling — In the Affect Labeling Condition, participants will be provided with instructions for how to verbalize their emotional response during the stressor.
  Arms: Affect Labelling Condition

SUMMARY:
Opioid use disorder is a major public health problem. Although there are effective treatments for this disorder, many people still relapse and thus there is a need for new treatments to improve outcomes. People who have a strong emotional and physical response to stress are at a higher risk of relapse. The goal of this project is to test the effect of strategies to reduce response to stress in people diagnosed with opioid use disorder. Men and women diagnosed with opioid use disorder will be recruited for a one-session study. Participants will be randomly assigned to one of three brief instructional conditions followed by a brief laboratory stress test. Investigators hypothesize that, compared to education about stress, brief strategies to help people cope with negative emotions will reduce responses to stress and increase tolerance of stress. If this hypothesis is supported, it will inform the development of new treatments to improve outcome in opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* primary diagnosis of opioid use disorder
* ability to read and provide informed consent

Exclusion Criteria:

* major psychiatric or medical condition that would interfere with the ability to complete study procedures
* current opioid withdrawal
* presence of another current substance use disorder at a severity requiring acute treatment
* endocrine disease or current steroid prescription
* opioid-positive urine drug screen or breath alcohol test on the data or enrollment (not including prescribed medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
In accordance with NIH policies for data sharing, data resulting from this project will be made available to qualified individuals within the scientific community. By data, this means the recorded, factual material necessary to document and support the research findings. Data will first be checked in accordance with the Data Safety and Monitoring Plan to ensure accuracy and completeness. To comply with pertinent local and federal regulations regarding the confidentiality of research data, any shared data would be free of identifiers that would permit linkage to research participants, and free of content that would create unacceptably high risks of subject identification. Data will be available to other researchers upon request to the study PI through a data sharing agreement after the primary paper has been accepted for publication in compliance with the NIH policy for the timely release and sharing of data.

REFERENCES:
- [Derived] McHugh RK, McCarthy MD, Bichon JA, Nguyen MD, Kneeland EK, Ellis RA, Dillon DG, Fitzmaurice GM. Effects of behavioral interventions on stress reactivity in adults with substance use disorders. Psychol Addict Behav. 2024 Dec;38(8):819-826. doi: 10.1037/adb0001032. Epub 2024 Sep 12. PMID 39264682
- [Derived] McHugh RK, Nguyen MD, Fitzmaurice GM, Dillon DG. Behavioral strategies to reduce stress reactivity in opioid use disorder: Study design. Health Psychol. 2020 Sep;39(9):806-814. doi: 10.1037/hea0000862. PMID 32833482

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psychoeducational Control | Affect Regulation Condition | Affect Labelling Condition
Started | 39 | 40 | 40
Completed | 39 | 40 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychoeducational Control | Affect Regulation Condition | Affect Labelling Condition | Total
Number analyzed (Participants) | 39 | 40 | 40 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.08 (11.79) | 43.83 (11.14) | 40.40 (10.0) | 41.87 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 12 | 40
  Male | 27 | 24 | 28 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4 | 8
  Not Hispanic or Latino | 34 | 39 | 36 | 109
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 31 | 36 | 34 | 101
  More than one race | 1 | 3 | 5 | 9
  Unknown or Not Reported | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Negative Affect
Description: Negative affect will be measured using the Negative Affect Subscale of the Positive and Negative Affect Schedule. This is a 10-item self-report measure on which respondents rate how strongly they are experiencing negative emotion. The range of scores is 10-50, with higher scores representing higher negative affect.
Time Frame: Change measured over 2 time points during this 1-session study experiment (from start of a stress induction task to completion; approximately 10-15 minutes).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Psychoeducational Control | Affect Regulation Condition | Affect Labelling Condition
Number analyzed (Participants) | 39 | 40 | 40
scores on a scale | 1.67 (8.70) | 1.25 (6.36) | 3.60 (6.93)

2. Primary Outcome: Distress Tolerance
Description: Distress tolerance will be measured using the Computerized Mirror Tracing Persistence Task. This is a computer-based task in which participants trace a mirror on the screen using the cursor. Participants are asked to persist at the task for as long as possible. Time to discontinuation is used as a measure of distress tolerance (in seconds). Longer duration reflects better tolerance of distress.
Time Frame: Time-to-event outcome; during this 1-session study, this will measure time to outcome (discontinuation of task) from time of initiation of the stress induction task up to a maximum of 15 minutes later.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Psychoeducational Control | Affect Regulation Condition | Affect Labelling Condition
Number analyzed (Participants) | 39 | 40 | 40
seconds | 244.72 (151.72) | 227.07 (169.48) | 217.34 (148.67)

3. Secondary Outcome: Change in Cortisol Response
Description: Cortisol levels will be measured using saliva samples. Salivary cortisol levels are measured on a continuous scale (micrograms/deciliter).
Time Frame: Change measured over 2 time points during this 1-session study (from start of stress induction task to 30 minutes after completion; approximately 40-45 minutes).
Population: Values more than 3 standard deviations from the mean were excluded.
Measure: Mean (Standard Deviation); unit: micrograms/deciliter
Arm/Group | Psychoeducational Control | Affect Regulation Condition | Affect Labelling Condition
Number analyzed (Participants) | 36 | 34 | 34
micrograms/deciliter | -0.07 (1.45) | -0.07 (1.02) | -0.63 (1.82)

4. Secondary Outcome: Change in Skin Conductance Level
Description: Skin conductance level is a physiological outcome that will be measured using electrodes placed on participants fingers, connected to a Biopac MP150 system with an ECG amplifier. Change will be measures by subtracting the maximum value during the stress task from the value at the end of a baseline recording.
Time Frame: Change measured over 2 time points during this 1-session study (prior to and during the stress induction task; approximately 10-15 minutes).
Population: Participants with data missing due to technical issues with data collection were excluded.
Measure: Mean (Standard Deviation); unit: microsiemens
Arm/Group | Psychoeducational Control | Affect Regulation Condition | Affect Labelling Condition
Number analyzed (Participants) | 30 | 26 | 29
microsiemens | 0.68 (1.12) | 0.80 (0.94) | 1.16 (1.21)

5. Secondary Outcome: Change in Opioid Craving
Description: Self-report of opioid craving will be measured using the Opioid Craving Scale, a 3-item measure, with a range of 0-30, with higher scores representing strong opioid craving.
Time Frame: Change measured over 2 time points during this 1-session study (immediately prior to and at the completion of the stress induction task; approximately 10-15 minutes).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychoeducational Control | Affect Regulation Condition | Affect Labelling Condition
Number analyzed (Participants) | 39 | 40 | 40
score on a scale | -0.26 (1.60) | -0.18 (1.57) | 0.60 (2.01)

ADVERSE EVENTS:
Time Frame: 1-3 hours (during the single-session study)
Arm/Group | Psychoeducational Control | Affect Regulation Condition | Affect Labelling Condition
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/39 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT03616379/Prot_SAP_000.pdf